CLINICAL TRIAL: NCT01411098
Title: A Phase I Dose-Intensification Study Using Radiation Therapy and Concurrent Cisplatin and Etoposide for Patients With Inoperable Non-small Cell Lung Cancer
Brief Title: Radiation Therapy, Cisplatin, and Etoposide in Treating Patients With Non-small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7506; NCI-2011-01752 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7506 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (radiation therapy and chemotherapy) (Experimental): Patients undergo 3D-CRT or IMRT 5 days a week for 8 weeks. Patients also receive cisplatin IV over 60 minutes on days 1, 8, 28, and 36 and etoposide IV over 60 minutes on days 1-5, and 28-32.
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy; Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy — Undergo 3D-CRT
  Other Names: 3D conformal radiation therapy; 3D-CRT
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213

SUMMARY:
This phase I trial studies the side effects and best dose of radiation therapy when given together with cisplatin and etoposide in treating patients with non-small cell lung cancer that cannot be removed by surgery. Radiation therapy uses high energy x rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Drugs, such as cisplatin, may make tumor cells more sensitive to radiation therapy. Giving radiation therapy together with cisplatin and etoposide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of escalating doses of radiotherapy (RT) administered concomitantly with a fixed dose of cisplatin and etoposide within the same overall treatment time.

OUTLINE: This is a dose-escalation study of radiation therapy.

Patients undergo 3-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiotherapy (IMRT) 5 days a week for 8 weeks. Patients also receive cisplatin intravenously (IV) over 60 minutes on days 1, 8, 28, and 36 and etoposide IV over 60 minutes on days 1-5 and 28-32.

After completion of study treatment, patients are followed up at 8 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed unresectable Stage IIB or Stage III non-small cell lung cancer of any histologic-subtype appropriate for definitive concurrent chemotherapy and radiation as determined by multi-disciplinary assessment; all detectable tumor should be encompassable by radiation therapy fields, including both the primary tumor and the involved regional lymph nodes
* Granulocytes >= 1500/ul
* Platelets >= 100,000/ul
* Bilirubin < 1.5 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) < 2 upper limit of normal (ULN)
* Creatinine clearance must be > 60ml/min
* Eastern Cooperative Oncology Group (ECOG) 0 to 1
* Weight loss =< 5% in the previous six months unless weight loss is intentional (per judgment of study medical doctor [MD])
* Forced expiratory volume in one second (FEV1) must be >= 1.0 L
* Patients must sign a study-specific informed consent form prior to study entry
* Patients must have measurable disease on the 3D planning computed tomography (CT)
* Patient must have a completed 3D plan and the attending physician must have reviewed and approved the dose volume histograms as follows: total lung volume percentage receiving at least 20 Gy (V20) =< 35%, and mean lung dose =< 20 Gy

Exclusion Criteria:

* Mixed histology or undifferentiated small cell carcinoma, any stage
* Concurrent malignancy except non-melanomatous skin cancer or prior cancer if disease-free for one year or more
* Patients with malignant pleural effusions or significant pericardial effusions
* Pregnant or lactating females
* Severe neuropathy greater than or equal to grade 2
* Severe sensorineural hearing loss greater or equal to grade 2
* No clinically significant history of cardiac disease, (i.e. uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the past year, or cardiac ventricular arrhythmias requiring medication)
* Any significant or severe medical conditions or psychiatric or social conditions that would preclude adherence to the protocol or compliance with study treatments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
MTD of radiotherapy, in terms of number of daily fractions, that can be delivered using 3D-CRT or IMRT with the standard cisplatin/etoposide regimen | Up to 8 weeks after completion of radiotherapy
  The MTD will be the highest dose at which no more than one of six patients experience a dose-limiting toxicity. Toxicity will be scored using the National Cancer Institute Common Toxicity Criteria version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpen Patel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States